CLINICAL TRIAL: NCT00864188
Title: Phase 1 The Influence of Probiotics in a Drinkable Yogurt on Skin Health
Brief Title: The Influence of Probiotics in a Drinkable Yogurt on Skin Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 08.29.NRC
Record Dates: First submitted 2009-03-13; First posted 2009-03-18 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2009-09

CONDITIONS: Skin Health
Keywords: skin health; probiotics; dairy; oral
MeSH Terms: interventions — L 644711; beta Carotene; Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): Glucono-Delta-Lactone acidified milk containing no bacterial strains
  Interventions: Dietary Supplement: no bacterial strains
- 2 (Experimental): Glucono-Delta-Lactone acidified milk containing one probiotic strain called Lactobacillus paracasei NCC2461.
  Interventions: Dietary Supplement: One probiotic strain - Lactobacillus paracasei NCC2461
- 3 (Placebo Comparator): Fermented milk containing two standard bacterial strains for acidification - Streptococcus thermophilus and Lactobacillus delbrueckii subsp.bulgaricus.
  Interventions: Dietary Supplement: Two standard yogurt fermenting bacterial strains - Streptococcus thermophilus and Lactobacillus delbrueckii subsp. bulgaricus
- 4 (Experimental): Fermented milk containing two standard bacterial strains for acidification - Streptococcus thermophilus and Lactobacillus delbrueckii and one probiotic strain called Lactobacillus paracasei NCC2461.
  Interventions: Dietary Supplement: One probiotic strain - Lactobacillus paracasei NCC2461; Dietary Supplement: Two standard yogurt fermenting bacterial strains - Streptococcus thermophilus and Lactobacillus delbrueckii subsp. bulgaricus
- 5 (Experimental): Fermented milk containing two standard bacterial strains for acidification - Streptococcus thermophilus and Lactobacillus delbrueckii, one probiotic strain called Lactobacillus paracasei NCC2461 and Vitamin B2,B3, C and E, Beta Carotene and an Oil.
  Interventions: Dietary Supplement: One probiotic strain - Lactobacillus paracasei NCC2461; Dietary Supplement: Two standard yogurt fermenting bacterial strains - Streptococcus thermophilus and Lactobacillus delbrueckii subsp. bulgaricus; Dietary Supplement: Vit B2, B3, C and E, Beta Carotene and Oil

INTERVENTIONS:
Dietary Supplement: no bacterial strains — Glucono-Delta-Lactone acidified milk containing no bacterial strains
  Arms: 1
Dietary Supplement: One probiotic strain - Lactobacillus paracasei NCC2461 — Glucono-Delta-Lactone acidified or fermented milk containing one probiotic strain.
  Arms: 2; 4; 5
Dietary Supplement: Two standard yogurt fermenting bacterial strains - Streptococcus thermophilus and Lactobacillus delbrueckii subsp. bulgaricus — Fermented milk containing two standard yogurt bacterial strains.
  Arms: 3; 4; 5
Dietary Supplement: Vit B2, B3, C and E, Beta Carotene and Oil — Fermented milk containing nutritional supplements
  Arms: 5

SUMMARY:
The aim of this study is to test if probiotics administered to healthy female subjects in a dairy format have any skin health benefits.

DETAILED DESCRIPTION:
This is a placebo-controlled, double blind, randomized, single center, human clinical trial aimed at assessing the influence of probiotics on skin health in healthy female subjects, when administered in a food matrix over a period of 5 months.

It will consist of five groups(40 subjects/group). The first group (1) of subjects will receive acidified milk that does not contain bacterial strains. The second group (2) will receive acidified milk that contains one specific probiotic strain. The third group (3) will receive fermented milk that contains a standard mix of yogurt bacterial strains. The fourth group (4) will receive fermented milk, containing the same standard mix of yogurt bacterial strains as in group 3 plus the same specific probiotic strain as in group 2. Finally, the fifth group (5) will receive fermented milk, containing the same standard mix of yogurt bacterial strains as in group 3 and 4 plus the same specific probiotic strain as in group 2 and 4 plus a mix of antioxidants.

This study will address whether:

A.The bioefficacy of a specific probiotic strain is influenced by a milk matrix.

B.Whether other bacterial strains impact the bioefficacy of this specific probiotic strain, and validate whether or not the bioefficacy is related entirely to the activity of this specific probiotic strain.

C.Whether nutritional supplements impact the bioefficacy of a specific probiotic strain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women as assessed by medical history and standard medical examination
* Caucasian
* Age: 25-55 y (inclusive)
* Normal BMI ≤ 30
* Skin type 1-111
* Regular Hormonal Cycle
* Having given his/her written informed consent
* Willing to avoid the consumption of fermented dairy products
* Minimum consumption of dark chocolate during the period of the study

Exclusion Criteria:

* Smoker
* Pregnant or lactating women
* Post menopausal women
* Heavy alcohol intake (usually consuming more than 3 standard drinks/day)
* Intake of chronic medications except oral contraceptive
* Vitamin and/or mineral and/or antioxidant supplementation over the 3 months preceding the initiation of the study and throughout the study.
* Having skin cancer or genetic disposition to skin cancer
* Regular exposure to artificial UVR
* Daily exposure to sun more than one week over the 2 months preceding the initiation of the study
* Planned vacation to sun during the period of the study.
* Excessive tea drinkers (more than 2 cups a day of green or black tea).
* Excessive consumer of fermented dairy products (more than 150g per day).
* Excessive consumer of dark chocolate (> 25g per day).
* Regular high exercise such as a marathon
* Subject who regularly takes saunas (dry or wet) or swims daily.
* Subject who cannot be expected to comply with treatment
* Currently participating or having participated in another interventional clinical trial during the last 3 months prior to the beginning of this study.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss | baseline, 1 month, 2 months, 3 months, 5 months and 6 months

SECONDARY OUTCOMES:
Biopsy markers: transglutaminase, filagrin, involucrin, loricrin (mRNA) | baseline and at 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für umweltmedizinische Forschung (IUF) an der Heinrich-Heine-Universität Düsseldorf gGmbH, Düsseldorf, Germany